CLINICAL TRIAL: NCT02039362
Title: Prevention of Hepatitis B Virus (HBV) Mother-to-Child (MTC) Transmission by Serovaccination of Newborns and Use of Tenofovir DF During the Last Trimester of Pregnancy in Mothers With HBV DNA Above 100, 000 I.U/mL
Brief Title: Prevention of Hepatitis B Virus Vertical Transmission by Serovaccination and Tenofovir During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, Professor at Paris VII University (Denis Diderot), physician, Hopital Lariboisière
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Liver002
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy; HBV
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tenofovir (Other): tenofovir DF one pill (245 mg) per day from week 28 of pregnancy to week 12 after birth
  Interventions: Drug: Tenofovir DF

INTERVENTIONS:
Drug: Tenofovir DF — Tenofovir DF will be started at week 28 of pregnancy and stopped or not, according to the physician's decision, at week 12 after birth

SUMMARY:
The risk of vertical HBV transmission is related to HBV DNA level in pregnant women, around 30% in women with HBV DNA above 1, 000 000 I.U/mL despite serovaccination of newborns. Using tenofovir DF during the last trimester of pregnancy allows to reduce the risk, but data from Western countries are needed.

DETAILED DESCRIPTION:
The prevalence of HBs Ag carriage in pregnant women varies in France, according to the native country, with higher rates in those originating from sub-Saharan Africa and Asia (5 to 8% in Parisian area). The level of HBV DNA varies according to HBe status and geographical origin, and is strongly predictive of the risk of HBV mother-to-child transmission (MTCT). The rate of vertical transmission (Yuan J et al. J Viral Hepatitis 2006) was 0% in newborns to mothers with HBV DNA less than 100,000 copies/mL and up to more than 40% in newborns to mothers with HBV DNA above 8 Log10 copies/mL, despite serovaccination at birth, thus justifying the use of tenofovir DF during the last trimester of pregnancy in highly viraemic pregnant women, as mentionned in EASL 2012 Guidelines. Data are needed concerning the results of this strategy in western countries, justifying this prospective study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* positive for HBs Ag
* HBV DNA above 100,000 I.U/mL

Exclusion Criteria:

* HIV co-infection
* HDV co-infection
* requiring, according to the physician's decision, a treatment for herself and not only to prevent HBV MTC transmission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of chronically infected (positive HBs Ag) children born from mothers with HBV DNA above 100, 000 I.U/mL being given tenofovir during the last trimester of pregnancy. | At 9 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O SELLIER, MD, PhD, Principal Investigator — Hopital Lariboisiere, Paris, France
Locations (1):
- Hopital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sellier PO, Maylin S, Bercot B, Chopin D, Lopes A, Simoneau G, Evans J, Delcey V, Benifla JL, Simon F, Bergmann JF. Prospective interventional study of tenofovir in pregnancy to prevent vertical transmission of hepatitis B in highly viremic women. Eur J Gastroenterol Hepatol. 2017 Mar;29(3):259-263. doi: 10.1097/MEG.0000000000000793. PMID 27879486